CLINICAL TRIAL: NCT06114771
Title: The Evaluation of the Effect of Preoperatively Applied Throat Lozenges on Postoperative Sore Throat,Cough and Hoarseness in Patients Operated Under General Anesthesia in Oral and Maxillofacial Surgery Department
Brief Title: The Evaluation of the Effect of Preoperatively Applied Throat Lozenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Raha Akbarihamed, lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ank-Medipol-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Pain, Postoperative
Keywords: Pain; Anesthesia and Analgesia; Orthognathic Surgery
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orthognathic surgery patients / lozange (Active Comparator): Throat lozenge (strepsilis) was given to 30 patients,30 minutes before the operation (the dissolution rate of the lozenge was proven to be 6-9 minutes).
  Interventions: Other: strepsilis
- orthognathic surgery patients / candy (Placebo Comparator): Sugar dragee in the same size and shape was given to 30 patients 30 minutes before the operation. In order not to cause any complications, sugar patients were sucked and told not to chew.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: strepsilis — Throat lozenge (strepsilis) was given to patients 30 minutes before the operation (the dissolution rate of the lozenge was proven to be 6-9 minutes).
  Arms: orthognathic surgery patients / lozange
Other: Placebo — Sugar dragee in the same size and shape was given to 30 patients 30 minutes before the operation. In order not to cause any complications, sugar patients were sucked and told not to chew.
  Arms: orthognathic surgery patients / candy

SUMMARY:
Purpose:The aim of this study is to evaluate the effect of preoperative throat lozenge on pain relief in the postoperative period of the mucosal damage caused by intubation in patients who underwent operations in the head and neck region under general anesthesia.

Methods: 60 patients were included in this study who were hospitalized in the inpatient service of the Oral and Maxillofacial Surgery department, This study was single-blind and performed by the same practitioner. Throat lozenge (strepsilis) was given to patients 30 minutes before the operation (the dissolution rate of the lozenge was proven to be 6-9 minutes).The postoperative sore throat was evaluated by VAS scale (0=no pain, 10=unbearable pain), and cough and hoarseness were evaluated with a four-point Likert scale (0=absent, 3=severe) at 1, 4, 6, 12, and 24 hours.

DETAILED DESCRIPTION:
Before the operation, blood sugar, urea, creatinine, electrolytes, prothrombin time, active partial thromboplastin time, and liver enzyme levels were determined in all patients. Hemoglobin and hematocrit determinations were made. Electrocardiography and chest radiographs were taken. Patients whose biochemical tests were within normal limits were included in our study.

The study was single-blind and performed by the same practitioner. Throat lozenge (strepsilis) was given to 30 patients, and sugar dragee in the same size and shape was given to 30 patients 30 minutes before the operation (the dissolution rate of the lozenge was proven to be 6-9 minutes). In order not to cause any complications, sugar patients were sucked and told not to chew.

Before the initiation of general anesthesia, height, weight, intubation time, mallampati score and ASA classification, the name of the operation, the start and end time of the operation, smoking, tube number, and whether spasms occurred were recorded. Patients taken to the service in the postoperative period were rested by wearing an oxygen mask. Postoperative sore throat VAS scale (0 = no pain, 10 = unbearable pain), cough, and hoarseness were assessed at 1, 4, 6, 12, and 24 hours with a four-point Likert scale (0 = absent, 3 = severe).

ELIGIBILITY:
Inclusion Criteria:

Being over 18 years old Having ASA I and II scores Clinical diagnosis of Alzheimer's Disease Must be able to swallow tablets

Exclusion Criteria:

Being over 60 years old Complex intubation cases Insulin dependent diabetes Thyroid disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-08-06 (Actual)

PRIMARY OUTCOMES:
preoperatively applied Throat lozenges on postoperative Sore Throat,Cough and Hoarseness in patients operated under General Anesthesia | 1, 4, 6, 12, and 24 hours
  postoperatively; sore throat (POST)

CONTACTS AND LOCATIONS:
Overall Officials: mine CAMBAZOĞLU, Prof, Study Director — Ankara University faculity of Dentistry
Locations (1):
- Raha, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No